CLINICAL TRIAL: NCT06151041
Title: Microneedling Combined With Either Tranexamic Acid or PRP in Treatment of Pigmented Postacne Scars : A Split Face Comparative Study
Brief Title: Microneedling Combined With Either Tranexamic Acid or PRP in Treatment of Pigmented Postacne Scars
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham Youssef Mahmoud Moustafa, prof / Doaa samir sayed, Assiut University
Other Study IDs: post acne scars
Record Dates: First submitted 2023-05-26; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Pigmented Post Acne Scars

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the efficacy of Microneedling combined with Tranxemic acid compared with Micronedlling with PRP in treatment of Pigmented Post Acne Scars.

DETAILED DESCRIPTION:
Acne is a multifactorial chronic inflammatory disease of pilosebaceous unit, clinically characterised by the presence of comedones, inflammatory papules, pustules and sometimes nodules and cysts. It commonly occurs during adolescence and cause great psychological stress. Unfortunately, acne scarring is common and occurs easily in the course of the disease. It is one of the most common causes of facial scarring and treating acne scar is one of the most challenging cosmetic procedures . Patient with acne vulgaries is not only experience the primary inflammatory and non-inflammatory lesions, but also have secondary lesions such as scars, excoriations, post-inflammatory erythema, and dyspigmentation. Acne scars are pleomorphic and difficult to count or even photograph, and consensus concerning acne scar nomenclature and classification remains a matter of debate .

The pathophysiology driving acne scar development is attributed to an altered wound healing response initiated by cutaneous inflammation, leading to an imbalance in matrix degradation and collagen biosynthesis .

The ultimate severity is correlated with acne grade and delay in treatment of active disease . The end result is either an excess of collagen that manifests as hypertrophic/keloid scars or, more commonly, decreased collagen deposition that manifests as atrophic acne scars in 80 to 90 percent of cases.

Tranexamic acid (TXA); a plasmin inhibitor used to prevent fibrinolysis to reduce blood loss , is now gaining popularity as a depigmenting agent as it can block melanin synthesis in melanocytes by inhibiting plasmin-plasminogen system , as well as competitive-inhibition of tyrosinase activity due to its similarity to tyrosine structure .

Microneedling has been used to treat various dermatologic conditions, including scars, rhytides, and dyschromia . The treatment causes small channels of epidermal and dermal injury through the use of needles that puncture the skin . The damaged collagen is removed, and new growth and remodeling subsequently occur . The release of platelet-derived growth factors, fibroblasts, and elastic fiber formation contribute to neovascularization and neocollagenesis ..

Ultimately, this improves the appearance of scars, especially atrophic scars. Since microneedling minimally alters the epidermis, there are limited adverse effects and downtime compared to more invasive .

PRP consists of the patient's own plasma that is enriched with a concentration of platelets that exceeds normal levels. It also contains various growth factors, including platelet-derived growth factor (PDGF), transforming growth factor (TFG), vascular endothelial growth factor (VEGF), and insulin-like growth factor (IGF). These growth factors stimulate tissue remodeling and are associated with enhanced healing through the attraction of macrophages, upregulation of collagen synthesis, and promotion of tissue regeneration .

Microneedling has been known to be an effective treatment option for acne scars; however, the addition of PRP has only recently been investigated. The upregulation of growth factors associated with PRP is believed to augment the effects of microneedling to promote aesthetically superior tissue remodeling. Their synergistic effects offer a unique treatment approach .

ELIGIBILITY:
Inclusion Criteria:

1. - 40 Male or Female healthy patient with Pigmented facial acne scars.
2. - Age of patient 18 -35 years old .
3. - Co-operative patients .
4. - No history of allergy to traneximc acid .
5. - No history of bleeding disorder

Exclusion Criteria:

1. Presence of active Acne Lesions .
2. Patients having Keloid scaring and Keloid tendency .
3. History of bleeding disorder.
4. History of anticoagulant therapy.
5. Active Skin infection like Warts , Hereps , Bacterial infection .
6. Pregenancy and Lactation .
7. Patients below 18 years .
8. History of laser treatment or any other acne therapy within one month .
9. Use of any acne medication in oral and topical forms , including retiniods , antibiotics

Ages: 18 Years to 35 Years | Sex: All
Age Groups: Adult
Study Population: This split face comparative study included 40 patients , their ages ranging from 18-35 years old , Presented to our dermatological department and outpatient basis with the main complaint of post acne scars . The morphology of each scar must be assessed , and treatment designed according to the all types of scars , overall appearance and expectations of the patient. The patient must be adequately counseled that the goal of treatment is improvement rather than perfection , as deep scars cannot be entirely eliminated
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
To evaluate the comparison between the efficacy of Microneedling combined with Tranexmic acid on the right side of the face and efficacy of PRP on the left side of the face in treatment of pigmented post acne scars | 1 year
  To evaluate the comparison between the efficacy of Microneedling combined with Tranexmic acid on the right side of the face and efficacy of PRP on the left side of the face in treatment of pigmented post acne scars in 1 year and this evaluation can be measured by a Questionnaire throught study completion and take photograghes each session .

REFERENCES:
- [Background] Khunger N; IADVL Task Force. Standard guidelines of care for acne surgery. Indian J Dermatol Venereol Leprol. 2008 Jan;74 Suppl:S28-36. PMID 18688101
- [Background] Lee WJ, Jung HJ, Lim HJ, Jang YH, Lee SJ, Kim DW. Serial sections of atrophic acne scars help in the interpretation of microscopic findings and the selection of good therapeutic modalities. J Eur Acad Dermatol Venereol. 2013 May;27(5):643-6. doi: 10.1111/j.1468-3083.2011.04330.x. Epub 2011 Nov 5. PMID 22054253
- [Background] Layton AM, Henderson CA, Cunliffe WJ. A clinical evaluation of acne scarring and its incidence. Clin Exp Dermatol. 1994 Jul;19(4):303-8. doi: 10.1111/j.1365-2230.1994.tb01200.x. PMID 7955470